CLINICAL TRIAL: NCT07338006
Title: Comparative Outcomes of Chest Wall Reconstruction Using Twisted Steel Wires Versus Bone Cement: A Cohort Study
Brief Title: Chest Wall Reconstruction Cohort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Doctor, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2025/1719/SIMS
Record Dates: First submitted 2026-01-03; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Chest Wall Tumor; Reconstructive Surgical Procedure; Malignancy
Keywords: Chest wall reconstruction; Bone cement; Stainless steel wire; Thoracic surgery; Postoperative pain; Functional outcomes
MeSH Terms: conditions — Neoplasms; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bone cement Arm (Active Comparator): This arm included patients that underwent chest wall reconstruction using bone cement
  Interventions: Procedure: chest wall reconstruction
- Steel wire arm (Experimental): This arm included patients that underwent chest wall reconstruction with steel wires
  Interventions: Procedure: Chest wall reconstruction

INTERVENTIONS:
Procedure: chest wall reconstruction — Chest wall reconstruction was performed using PMMA bone cement molded intraoperatively over a polypropylene mesh to form a rigid prosthesis. The construct was fixed to the adjacent ribs with nonabsorbable sutures or wires.
  Arms: Bone cement Arm
Procedure: Chest wall reconstruction — chest wall reconstruction was achieved using twisted stainless steel wires (No. 05) anchored to the adjacent ribs or sternum, creating a flexible rib framework. The wires were tightened in a crisscross fashion to provide stable yet dynamic support.
  Arms: Steel wire arm

SUMMARY:
Chest wall reconstruction following tumor or infection-related resections remains a challenging aspect of thoracic surgery, requiring restoration of structural stability and preservation of respiratory mechanics. While polymethyl methacrylate (PMMA) bone cement has long been used for rigid reconstruction, its limitations-including high cost, rigidity, infection risk, and interference with normal respiratory motion-pose challenges in resource-constrained settings. Twisted stainless steel wires offer a low-cost, flexible alternative that allows dynamic chest wall movement and easier adaptability in low- and middle-income countries such as Pakistan.

To compare postoperative outcomes, complications, and cost-effectiveness of chest wall reconstruction using twisted stainless steel wires versus PMMA bone cement over a two-year period (January 2025 - December 2026).

This prospective cohort study was conducted in the Department of Thoracic Surgery, Services Hospital, Lahore, a high-volume tertiary care and referral center. Patients undergoing chest wall reconstruction following resection for tumors, infections, or trauma were enrolled and divided into two groups based on the reconstruction technique used: Group A (twisted steel wires) and Group B (PMMA bone cement). Parameters assessed included postoperative pain (VAS scores), respiratory function, chest wall stability, complications (infection, wound dehiscence, prosthesis exposure), duration of hospital stay, readmission rate, and cost of reconstruction. Data were analyzed to compare clinical and functional outcomes between both cohorts.

DETAILED DESCRIPTION:
Chest wall resection for tumors results in complex structural defects that require meticulous reconstruction to restore stability, protection, and respiratory function. The chest wall, composed of a combination of bony and soft tissue components, plays a crucial role in ventilation; thus, its reconstruction must achieve mechanical integrity while preserving physiologic mobility and minimizing postoperative morbidity.

Multiple techniques and materials have been developed for chest wall reconstruction, including synthetic meshes, titanium plates, and polymethyl methacrylate (PMMA) bone cement. PMMA remains widely used due to its moldability and compressive strength; however, its rigidity, low tensile strength, poor adhesion, and potential for thermal necrosis and infection limit its functional and clinical effectiveness. Furthermore, its high cost and non-dynamic properties make it less suitable in resource-constrained settings.

In contrast, twisted stainless steel wires (No. 05) offer a simple, durable, and cost-effective alternative. These wires provide robust mechanical support with dynamic flexibility, preserving normal respiratory motion and chest wall recoil. Recent advancements have demonstrated that wire-reinforced neorib configurations can achieve both tensile and compressive strength comparable to rigid prosthetics, while avoiding the static limitations of PMMA. Their affordability and availability make them particularly advantageous in low- and middle-income countries where economic feasibility dictates surgical decisions.

Recent studies have further explored biologic and synthetic prosthetic materials, microvascular flaps, and hybrid "biosandwich" techniques to optimize chest wall reconstruction outcomes. Nevertheless, data comparing simple, low-cost methods such as twisted steel wire constructs and PMMA-based reconstructions remain limited, particularly in regions with restricted access to advanced materials. In Pakistan, evidence is largely confined to isolated case reports, including a novel reconstruction of a neosternum using steel wires for recurrent sternal chondrosarcoma.

The present cohort study, conducted in the Department of Thoracic Surgery at Services Hospital, Lahore, aims to compare the outcomes of chest wall reconstruction using twisted stainless steel wires versus PMMA bone cement over two years from January 2025 to December 2026. By evaluating postoperative pain, respiratory function, chest wall recoil, and complication rates, this study seeks to provide evidence-based recommendations for the optimal reconstructive strategy in resource-limited healthcare environments.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years undergoing partial or full-thickness chest wall resection.
* Defects requiring rigid or semi-rigid reconstruction involving two or more ribs or the sternum.

Exclusion Criteria:

* Patients with small defects managed by primary closure or soft tissue-only reconstruction.
* Patients with concurrent major intrathoracic resections (e.g., pneumonectomy) may confound postoperative respiratory assessment.
* Recurrent disease requiring revision reconstruction.
* Patients unwilling or unable to provide consent or comply with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Assessment: | 24 hours, 48 hours and 7 days post-operatively
  Postoperative analgesia followed a standardized multimodal protocol of intravenous paracetamol and NSAIDs unless contraindicated, supplemented with intravenous morphine (0.05-0.1 mg/kg) as required. Thoracic epidural or paravertebral blockade was used selectively based on resection extent or anesthetist preference. Rescue analgesia was administered when VAS pain scores were ≥4 at rest or ≥5 during movement.

SECONDARY OUTCOMES:
Chest Wall Movement | 1 month and 3 months post-operatively
  Chest wall function was evaluated clinically at discharge, at 1-month follow-up, and at 3-month follow-up by the operating surgeon or thoracic fellow, and patients who underwent surgery earlier in the study period remain under active surveillance, providing a total follow-up duration of up to two years. Assessment included inspection for paradoxical movement during quiet and deep breathing and measurement of axillary excursion when feasible. Normal chest movement was defined as symmetrical expansion or ≥3 cm axillary excursion. Restricted movement was defined as <3 cm excursion, ≥25% asymmetry relative to the contralateral side, or patient-reported limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital, Lahore, Lahore, Punjab Province, Pakistan